CLINICAL TRIAL: NCT03704701
Title: The Interrogation of the Cardiomyopathy of Chronic Kidney Disease With advancEd caRdiac Imaging
Acronym: TICKER
Status: Terminated | Type: Observational
Why Stopped: COVID-19 pandemic; pre-pandemic recruitment sufficient for scientific validity
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN17RE700; 243630 (Other: Integrated Research Application System (IRAS) ID)
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases; Cardiomyopathies; Cardiovascular Diseases; Cardiac Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiomyopathies; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for routine clinical parameters and novel biomarkers of cardiovascular disease and fibrosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cardiac MRI and contrast-enhanced cardiac CT — Cardiac MRI Contrast-enhanced cardiac CT

SUMMARY:
Patients with kidney failure have a much higher risk of heart disease compared to people of the same age without kidney failure. The reason for this is not fully understood. In this project we will use Cardiac MRI (CMR), which is a very detailed scan of the heart and blood vessels, to try to better understand the cardiovascular changes that occur in kidney failure. We will perform CMR scans in 30 patients before and after dialysis (a treatment for patients with kidney failure) to see whether dialysis changes the heart muscle. The same patients will also undergo another type of heart scan, called a CT scan. This will allow us to compare the pictures from the 2 different types of scan to help us better understand any damage to the heart muscle that is present. Finally, we will test a new way to measure hardening of blood vessels on CMR. These three studies will help us to better understand the heart and blood vessel changes that happen in kidney failure. This research will also be useful for patients without kidney failure. We hope to be able to use it in the future to see which new treatments might be able to reduce the risk of heart disease in patients with kidney failure.

DETAILED DESCRIPTION:
Background: Patients with chronic kidney disease (CKD) are at a dramatically increased risk of cardiovascular disease. This risk is greatest in patients on dialysis and is not explained by conventional cardiovascular risk factors. Myocardial fibrosis, so called Cardiomyopathy of CKD (CM-CKD), in conjunction with excessive arterial calcification, forms the pathological basis for this excess risk. Due to limitations of using myocardial biopsy, combined with the inability to use gadolinium-enhanced imaging in patients with advanced CKD, there is an urgent need for reliable non-invasive ways of diagnosing and investigating CM-CKD.

Study participants: Adult patients established on regular hospital-based haemodialysis, with evidence of recurrent fluid overload requiring fluid removal by ultrafiltration on dialysis.

Study design: This is a single centre observational study. We will perform cardiac MRI (CMR), contrast CT and blood tests in 30 patients before haemodialysis, with a repeat CMR and blood tests post-dialysis.

Objectives: To assess:

1. If myocardial native T1 mapping on CMR is affected by fluid status and therefore test the validity of T1 mapping as a marker of fibrosis within the dialysis population?
2. If contrast-enhanced dynamic-equilibrium CT can refine insights into the myocardium in CM-CKD?
3. If novel CMR methods can effectively identify and delineate arterial calcification compared to CT?

Relevance: This project will have immediate clinical relevance by clarifying key questions in the diagnosis and investigation of CM-CKD. It will also inform as to the potential role for these novel imaging biomarkers as surrogate end-points for use in future clinical trials exploring disease specific drug therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-100 years at time of recruitment.
2. Established on regular day-time, hospital-based haemodialysis for >6 months.
3. History of recurrent fluid overload, defined as a mean of >1.5 litres fluid removal per dialysis session from an average of 3 consecutive sessions.
4. No previous clinical diagnosis of heart failure, or if previous clinical diagnosis of heart failure then must have preserved left ventricular function (ejection fraction >50% or reported as 'normal' or (similar)) on most recent transthoracic echo.
5. Ability to comply with study procedures, including ability to lie flat for up to 1 hour.
6. Ability to give informed consent.

Exclusion Criteria:

1. Standard contra-indications to MRI, including the presence of certain metallic objects in the body (e.g. non-MRI compatible cardiac devices, previous cranial surgery with ferromagnetic clips, metal fragments in eye, etc.) and severe claustrophobia.
2. Known allergy to iodinated radiological contrast.
3. Asthma (unless previous CT with contrast administration within the past 12 months without adverse effect).
4. Pregnancy, lactation or women of child-bearing potential not willing to use highly effective contraception for the duration of the study.
5. Any other reason considered by a study physician to make the subject inappropriate for inclusion.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients established on regular hospital-based haemodialysis, with evidence of recurrent fluid overload requiring fluid removal by ultrafiltration on dialysis.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Part 1A: Myocardial native T1 in response to changing fluid status | 24 hours
  Change in myocardial native T1 mapping (MOLLI) on cardiac MRI at visit 2, compared to visit 1, following removal of excess fluid by ultrafiltration.
Part 1B: Measurement of myocardial extracellular volume by CT (ECV-CT) | Baseline
  Comparison between myocardial extracellular volume on contrast-enhanced CT and myocardial native T1 times measured on cardiac MRI.
Part 1C: Vascular calcification on MRI | Baseline
  Comparison between Cardiac MRI and CT to detect the presence or absence of vascular calcification within the thoracic aorta at the level of the right pulmonary artery (PA).

CONTACTS AND LOCATIONS:
Overall Officials: Alastair J Rankin, MBChB, Principal Investigator — University of Glasgow
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided